CLINICAL TRIAL: NCT02198066
Title: A Comparison of Post-Sternotomy Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: DeRoyal Industries, Inc. (Industry); Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CC-2014-1
Record Dates: First submitted 2014-03-27; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-03

CONDITIONS: Impaired Wound Healing; Postoperative Wound Infection-deep
Keywords: Sternotomy incision; Silver dressing; Sternal wound infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dry Sterile Dressing (Other): Subjects in this study arm received a dry sterile dressing (Primapore®, Smith & Nephew), a one-piece, peel-and-stick, non-transparent dressing. This dressing is the standard of care at the study facility for this population and was left in place for either 24 to 48 hours.
  Interventions: Other: Dry Sterile Dressing
- Metallic Silver Dressing (Active Comparator): Subjects in this arm received a metallic silver dressing (Acticoat Post-Op®, Smith & Nephew), a one-piece, peel-and-stick and non-transparent dressing. This dressing is an absorbent postoperative dressing consisting of a nanocrystalline silver-coated polyurethane layer, a white polyurethane foam and an adhesive coated waterproof polyurethane film layer. Acticoat Post-Op may be left in place over a wound for up to 7 days. The manufacturers note that the product should not be used in patients with known silver allergies and that it may cause transient discoloration of the skin.
  Interventions: Other: Metallic Silver Dressing
- Ionic Silver Dressing (Active Comparator): Subjects in this arm received an ionic silver dressing (Dermanet Ag®, DeRoyal), a semi-transparent dressing that includes silver, alginate, and maltodextrin. The dressing was cut to fit the incision and then covered with a transparent dressing (Transseal®, DeRoyal). This dressing should not be used on patients with known sensitivity to alginates (a seaweed based component).
  Interventions: Other: Ionic Silver Dressing

INTERVENTIONS:
Other: Dry Sterile Dressing — Described in Arm Description.
  Other Names: Primapore (Smith & Nephew)
  Arms: Dry Sterile Dressing
Other: Metallic Silver Dressing — Described in Arm Description.
  Other Names: Acticoat Post-Op (Smith & Nephew)
  Arms: Metallic Silver Dressing
Other: Ionic Silver Dressing — Described in Arm Description.
  Other Names: Dermanet (DeRoyal)
  Arms: Ionic Silver Dressing

SUMMARY:
The purpose of this study was to determine which of three types of dressings, a dry sterile dressing, a metallic silver dressing or an ionic silver dressing provided better patient outcomes for the post-sternotomy cardiac surgery patient population. In this prospective, randomized controlled trial, the hypothesis was that subjects who received either of the silver impregnated dressings would have better outcomes (better wound healing, less discomfort, and less incidence of infection). Investigators also evaluated dressing factors such as adherence, time for application and ease of use.

DETAILED DESCRIPTION:
No other information included.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 21 years of age) inpatients awaiting cardiac surgery or outpatients seen in the pre-surgical testing area prior to admission for surgery
* Having surgery at the study setting
* English-speaking
* Able to understand and give consent
* Had the approval of their cardiothoracic surgeon to participate
* Had no known sensitivity to silver
* Had no known sensitivity to alginates

Exclusion Criteria:

* Known sensitivity to silver
* Known sensitivity to alginates

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2010-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Wound Healing | 5 days postoperatively or day of discharge, whichever came first
  The primary outcome measure in this study was wound healing, defined as the degree of wound approximation, skin integrity, exudate, and presence/absence of necrotic tissue, assessed at postoperative day 5 or day of discharge. Wound approximation was assessed as total, partial (less than 2 centimeters of superficial separation), moderate (greater than 2 centimeters of superficial separation), or dehisced (complete separation of layers). Skin integrity was evaluated as normal (pink, no redness), inflamed, (heat, redness, swelling), or macerated within a 2.5 centimeter border of the incision. Exudate quality was assessed as purulent, blood, serosanguinous, or serous. Presence or absence of necrotic tissue was noted.

SECONDARY OUTCOMES:
Patient Comfort | 5 days postoperatively or day of hospital discharge, whichever came first
  The secondary outcome measure in this study was patient comfort with the dressing in place and upon removal. Comfort was measured using a 0-10 scale, with 0 signifying no pain and 10 signifying maximum pain.

OTHER OUTCOMES:
Dressing Factors | 5 days postoperatively or at day of discharge, whichever came first
  Dressing factors of ease of application, removal, and incision assessment were measured on a 5-point Likert-type scale (1=very easy, 2=moderately easy, 3=neither easy nor hard, 4=moderately hard, and 5=very hard). Dressing integrity was assessed as suture line exposed, poorly sealed (imperfect covering of the suture line with the potential for organism entry), or well-sealed.
Sternal Wound Infection | 30 days postoperatively
  Investigators evaluated sternal wound infection presence and type (superficial or deep) using Centers for Disease Control/National Healthcare Safety Network surveillance definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy D. Jennings, DNP, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States